CLINICAL TRIAL: NCT03411330
Title: Safety and Efficacy of Addition of Hyaluronidase to Lidocaine and Bupivacaine in Scalp Nerves Block in Elective Craniotomy Operations, Comparative Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Mohamed, Ahmed A., M.D. (Individual); Tarek Ahmed Radwan (Unknown); Mohamed Mahmoud Mohamed (Unknown); Hatem Abdellatif Mohamed (Unknown); Badawy Mohammed Al-Kholy (Unknown)
Responsible Party: Principal Investigator, Ahmed Abdalla, Assistant Professor of Anesthesia&I.C.U and Pain Clinic, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N-58/2017
Record Dates: First submitted 2017-12-27; First posted 2018-01-26 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Addition of Hyalase to Local Anesthetic in Scalp Block
MeSH Terms: interventions — Hyaluronoglucosaminidase; Lidocaine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: The investigators hypothesize that, the addition of hyaluronidase may affect the quality of the block by enhancing the spread of the local anaesthetics through the facial planes and thus, reaching the target nerves more easily, rapid and effective that may provide better effective block in short duration and lasting for longer duration. This effect will be measured in terms of "stress response" and " analgesic quality" Total sample size of 64 patients randomly allocated into two equal groups. According to study "Hyaluronidase in sub-Tenon's anesthesia for phacoemulsification" that was done and published in International Journal of Ophthalmology (2012) to detect difference in post-operative pain between those patients receiving Lidocaine only versus Lidocaine and hyaluronidase, sample size of 29 patients per group is needed with confidence level 95% power of the study 80% & type I error 0.05. Sample size calculation was done using Medcalc Software version 15.4.
Who Masked: Participant, Investigator
Masking Description: Prospective randomized double blinded clinical study on humans
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group H (Hyaluronidase added to local anaesthetics) (Active Comparator): group H scalp block will be done using lidocaine (2%) in a maximum dose of 300 mg and bupivacaine (0.5%) with maximum allowed dose 175 mg , Hyaluronidase will be added in in a dose of 1500 IU . The scalp block technique includes infiltrating local anaesthetic to 7 nerves on either side. This is an anatomical block and not just a ring block. At the end of the scalp block further local anesthetic can be infiltrated locally to the pin sites and 7 nernes supraorbital nerve, a branch of the trigeminal nerve,supratrochlear nerve, a branch of the trigeminal nerve.
  zygomaticotemporal nerve,auriculotemporal nerve, lesser occipital nerve, greater occipital nerve and greater auricular nerve
  Interventions: Drug: Hyaluronidase; Drug: Lidocaine; Drug: Bupivacaine
- Group A (local anaesthetics alone) (Active Comparator): Group A :scalp nerves block will be done using lidocaine (2%) in a maximum dose of 300 mg and bupivacaine (0.5%) with maximum dose of 175 mg The scalp block technique includes infiltrating local anaesthetic to 7 nerves on either side. This is an anatomical block, and not just a ring block. At the end of the scalp block; further local anesthetic can be infiltrated locally to the pin sites and 7 nernes Supraorbital nerve, a branch of the trigeminal nerve.
  supratrochlear nerve, a branch of the trigeminal nerve. zygomaticotemporal nerve, auriculotemporal nerve, lesser occipital nerve, greater occipital nerve, greater auricular nerve
  Interventions: Drug: Lidocaine; Drug: Bupivacaine

INTERVENTIONS:
Drug: Hyaluronidase — Scalp nerves block will be done using lidocaine (2%) in a maximum dose of 300 mg and bupivacaine (0.5%) with maximum allowed dose 175 mg in group A, Hyaluronidase will be added in group H in a dose of 1500 IU (The minimum and maximum effective doses of hyaluronidase are not known. The doses used range from0.75 IU/ml to 300 IU/ml
  Other Names: Hyaluronidase with lidocaine and bupivacaine
  Arms: Group H (Hyaluronidase added to local anaesthetics)
Drug: Lidocaine — lidocaine (2%) in a maximum dose of 300 mg and bupivacaine (0.5%)
  Other Names: Lidocaine alone
Drug: Bupivacaine — bupivacaine (0.5%)
  Other Names: Bupivacaine alone

SUMMARY:
Safety and efficacy of addition of hyaluronidase to lidocaine and bupivacaine in scalp nerves block in elective craniotomy operations,Comparative study

DETAILED DESCRIPTION:
Patients undergoing craniotomy operations are susceptible to many injurious stimuli such as skin incision, insertion of cranial pins, dural incision, dural and skin closure. They cause different levels of nociception and these stimuli can result in sudden increases in blood pressure and heart rate due to triggering stress response.

Strategies to blunt these noxious stimuli and attenuate this stress response include administration of systemic opioids, deepening the level of anaesthesia. Scalp nerves block by local anaesthetics also can be used.

However, most systemically administered medications studied for post-craniotomy pain usually associated with side effects such as sedation, nausea, and vomiting and depressed ventilation such events are particularly important for post-craniotomy patients.

Using regional aesthetic techniques in addition to general anaesthesia have been conducted as multimodality managements for post-craniotomy pain and to decrease systemic administration of analgesics and hence decrease their systemic complications.

The stress response is the hormonal and metabolic changes that follow injury or trauma. This includes wide range of endocrinological and immunological effects. The stress response to surgery is characterized by increased secretion of pituitary hormones and activation of the sympathetic nervous system. Hypothalamic activation of the sympathetic autonomic nervous system results in increased secretion of catecholamines from the adrenal medulla and release of norepinephrine from presynaptic nerve terminals. IL-6 is produced in substantial quantities at the site of a surgical wound.IL-6 enters the circulation, and its concentration correlates with the severity of surgery and thus with the magnitude of the tissue injury. At 24 to 36 h after surgery, the levels of IL-6 in the plasma reach preoperative values, because its production is attenuated. Postoperative pain behaves like wound on plasma IL-6: intense postoperative pain correlates with the magnitude of tissue injury and subsides days after. Pain in the first 24 hours after brain surgery is a significant problem, with 60% to 80% of patients experiencing moderate to severe pain.

Blockade of scalp innervation which anesthetises both the superficial and deep layers of the scalp, was used as a means of decreasing hemodynamic reactions during and after craniotomy operations. Various protocols to control postoperative pain were suggested, including infiltration of the scalp with local anaesthetics. These include the use of 0.5% bupivacaine combined with additional lidocaine 2 %.

Hyaluronidase is a naturally produced enzyme, it's produced by various types of bacteria, and primary helps bacteria to dissolve hyaluronic acid that constitutes major component of the connective tissue substance thus helping spread of other bacterial products. On December 2005, the FDA approved a synthetic (recombinant or rDNA) human hyaluronidase. The addition of hyaluronidase to local anaesthetics has been shown to enhance safely and effectively the diffusion of the drug, thereby increasing the analgesic efficacy especially in the first minutes after injection

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ι and II.
2. Both males and females, age (18-60) years.
3. Supine position.
4. Glasco coma scale more than 12.
5. Elective craniotomy operations.

Exclusion Criteria:

1. ASA ΙII or IV
2. History of allergy to the study drugs.
3. Surgery to remove pituitary tumours or affecting pituitary hormones.
4. Glasco coma scale less than 12.
5. The need for postoperative ventilation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2018-04-22 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Post-operative pain evaluation | up to 24 hours postoperatively
  Post-operative VAS for pain post-operative.

SECONDARY OUTCOMES:
Haemodynamic Measures | Every 5 minutes during operation In first 24 hours postoperatively
  Effects on haemodynamics: Heart rate"beats per minute" intra and post-operative in both groups
Interleukin 6 measurement | Interleukin 6 level will be measured before surgery (9:00 A.M),30 minutes after scalp nerves block, 60 minutes after skin incision and after 6 hours post-operative.
  Measurement of level of interleukin 6 as an indicator of inflammatory response and pain
Intraoperative rescue dose of opioid | 6 hours postoperative then every 2 hours for 24 hours.
  Number of patients requiring intraoperative rescue doses of opioids
Time of first analgesic request | Intraoperative
  First time to seek analgesia (time of first analgesic request)
Haemodynamic effects | up to 24 hours postoperatively
  Effects on haemodynamics:, systolic, diastolic and mean arterial blood pressure" mm Hg".

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Via scholar Gate

REFERENCES:
- [Derived] Mohamed AA, Radwan TA, Mohamed MM, Mohamed HA, Mohamed Elemady MF, Osman SH, Safan TF, Khair TM, Ali NA, Fahmy RS, Belita MI, Abdalla SR, Seleem AA, Atta EM, Zaid OI, Ragab AS, Salem AE, AlKholy BM. Safety and efficacy of addition of hyaluronidase to a mixture of lidocaine and bupivacaine in scalp nerves block in elective craniotomy operations; comparative study. BMC Anesthesiol. 2018 Sep 15;18(1):129. doi: 10.1186/s12871-018-0590-9. PMID 30219027